CLINICAL TRIAL: NCT00977418
Title: Brain & Cognitive Changes After Reasoning or Physical Training in Cognitively Normal Seniors
Brief Title: Brain and Cognitive Changes After Reasoning or Physical Training in Cognitively Normal Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07-19; NIH 1RC1AG035954-01
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2012-06

CONDITIONS: Hearing Impaired
Keywords: Healthy Aging; Exercise; Cognition; Cognitive Training; Keeping healthy seniors as mentally efficient as possible
MeSH Terms: conditions — Hearing Loss; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No intervention (No Intervention): Seniors undergo all testing but remain current lifestyle
- Training (Experimental): Groups will undergo either physical or mental training. Physical training is 1 hour aerobic training 3 times per week for 12 weeks. Mental training is 1 hour Strategic Memory Advanced Reasoning Training 3 times per week.
  Interventions: Behavioral: SMART- Strategic Memory and Reasoning Training; Other: Physical Exercise

INTERVENTIONS:
Behavioral: SMART- Strategic Memory and Reasoning Training — Teach people to filter out un necessary or unimportant details to enhance mental efficiency. This training will be done over 12 weeks for 3 hours each week.
  Arms: Training
Other: Physical Exercise — The group with undergo 1 hour of aerobic exercise (at 50-70 % of the participants max oxygen intake) 3 times a week for 12 weeks.
  Arms: Training

SUMMARY:
Seniors 65 years of age and older represent one of the fastest growing segments of society with the population doubling within the next 25 years with dramatic rates of mental decline, costing society billions of dollars each year. The proposed research seeks to discover whether relatively short term mental or physical training can enhance gist reasoning, generalize to untrained cognitive areas and modify/strengthen brain function in areas susceptible to aging processes. To identify neuroprotective and non-pharmacological interventions to prevent mental decline and maximize cognitive brain health during the course of the adult lifespan has major public policy implications.

DETAILED DESCRIPTION:
Background: A significant potential exists to modify the structure and function of the aging human brain given intensive mental stimulation and physical activity. Age-related cognitive decline has consistently been identified on frontal lobe measures of executive control such as reasoning. Concomitantly, a greater vulnerability of frontal brain networks, which subserve executive control functions, has also been identified with aging. Preliminary evidence highlights the potential of reasoning training as well as physical training to modify and strengthen brain and cognitive function in seniors. Evidence from our lab indicates that frontally mediated, gist-based reasoning (defined as the ability to combine detail information to construct abstract meanings) offers a promising cognitive domain to train. Extracting gist meaning from the massive amount of incoming information is one of the most vital mental skills a healthy mind achieves. Purpose: This proposal is an innovative study to obtain data regarding the benefits of a (a) novel gist-based reasoning training program or (b) physical training on frontal-lobe mediated cognitive measures of executive control in cognitively normal seniors. The project will also employ newly developed (a) brain measures to chart changes in brain blood flow and connectivity combined with (b) a cognitive activation task specifically designed to measure brain regions engaged in gist reasoning versus detail processing. The project also examines shorter dose effects, i.e. after 6 weeks and 12 weeks, than previously examined as well as individual differences based on high and low performers for gist and physical training. Methods: 60 cognitively normal seniors between the ages of 60 and 75 years will be recruited for study and randomized into 1 of 3 groups. Each group will consist of 20 participants each: a reasoning-trained, a physical-trained and a wait-listed control group. Participants will be comprehensively screened to insure they are cognitively normal. Prior to intervention, participants' baseline gist and detail processing ability, battery of cognitive functions and fitness measures will be obtained. Structural and functional brain measures will also be obtained. Participants will undergo 12 weeks of gist-based training or physical training with measurement at midpoint, 6 weeks of training, endpoint 12 weeks of training and 4 weeks after training is completed. Training effects will be measured behaviorally in trained areas (reasoning & physical) and untrained cognitive areas. Additionally, structural and functional brain imaging will measure changes in cerebral blood flow, global and regional brain volume, white matter tracts, efficiency, activation patterns, and blood oxygenation with a particular focus on changes to frontal regions. Significance: The current study seeks to discover neuroprotective, nonpharmacological interventions that could prevent mental decline and strengthen cognitive brain health in seniors, with possible societal savings of billions of dollars. This will be one of the first training studies to explore short-term intensive reasoning and physical training, each documented as pivotal to cognitive brain health with the potential to strengthen frontal regions against the losses associated with aging.

ELIGIBILITY:
Inclusion Criteria:

* The study will include 60 cognitively normal seniors between the ages of 60 and 75 years.
* Participants will have normal IQ, be native speakers of English and have a minimum of high school education.

Exclusion Criteria:

* Participants with a previous history of stroke, diabetes, untreated hypertension, major surgeries within the past 6 months, major psychiatric disorder, depression or cognitive impairment will be excluded.
* Additionally, anyone that has a condition that would exclude them from MRI will not be included.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cognitive Scores | begining (0 weeks), middle (6 weeks) and end (12 weeks) of study

SECONDARY OUTCOMES:
MRI images | begining (0 weeks), middle (6 weeks) and end (12 weeks) of study

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Chapman, Ph.D., Principal Investigator — The University of Texas at Dallas
Locations (1):
- The University of Texas at Dallas, Dallas, Texas, United States

REFERENCES:
- [Derived] Motes MA, Yezhuvath US, Aslan S, Spence JS, Rypma B, Chapman SB. Higher-order cognitive training effects on processing speed-related neural activity: a randomized trial. Neurobiol Aging. 2018 Feb;62:72-81. doi: 10.1016/j.neurobiolaging.2017.10.003. Epub 2017 Oct 12. PMID 29121545